CLINICAL TRIAL: NCT06508255
Title: Time-restricted Eating and Cognition (ChronoBEAT)
Brief Title: Time-restricted Eating and Cognition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Prof. Dr. Olga Ramich (German Institute of Human Nutrition) (Unknown); Freie Universität Berlin (Other); German Center for Diabetes Research (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Soyoung Q Park, Prof. Dr. Soyoung Q Park (Principal Investigator), German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ChronoBEAT
Record Dates: First submitted 2024-05-30; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Time Restricted Eating; Intermittent Fasting
Keywords: Time-restricted eating; Time-restricted feeding; Cognition; Decision-making; Behaviour; Brain Activity; Food Intake; Diet; Microbiome; Sleep; Physical Activity
MeSH Terms: conditions — Intermittent Fasting; Behavior; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time-Restricted Eating (Experimental)
  Interventions: Behavioral: Early Time-Restricted Eating
- Late Time-Restricted Eating (Experimental)
  Interventions: Behavioral: Late Time-Restricted Eating

INTERVENTIONS:
Behavioral: Early Time-Restricted Eating — Eat between 8:00 and 16:00 for 2 weeks
  Other Names: early TRE; eTRE; eTRF
  Arms: Early Time-Restricted Eating
Behavioral: Late Time-Restricted Eating — Eat between 13:00 and 21:00 for 2 weeks
  Other Names: late TRE; lTRE; lTRF
  Arms: Late Time-Restricted Eating

SUMMARY:
This study aims to investigate how time-restricted eating (TRE), more specifically TRE at different times (early vs late in the day), influences brain activity, behavior, decision-making, food intake, physical activity, the gut microbiome and metabolic processes. The study intervention procedure is a replication of that described in Peters et al. (2021).

DETAILED DESCRIPTION:
This study aims to investigate the effects of different time-restricted eating (TRE) interventions on decision-making, brain activity and related processes in an all female cohort over 8 weeks. The study will have a within-subjects, randomised, crossover design, involving two TRE interventions with a comparable feeding and fasting window of 8:16h respectively- early TRE (eating window: 08:00-16:00) and late TRE (eating window: 13:00-21:00). After completing a screening visit, participants will complete a two-week observational phase in which they record their habitual food intake, as well as sleep and physical activity assessment. After this observational phase, participants will be randomly assigned to one of two study arms (early TRE/late TRE or late TRE/early TRE). Here they will complete both TRE interventions for two weeks each, separated by a washout phase of two weeks. During these phases they will record their food intake and physical activity and sleep will be assessed. The participants will be invited for 4 laboratory study visits during this time, at the beginning and end of each TRE intervention.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* legally competent
* physically and mentally healthy
* BMI: 19-35 kg/m²
* fluent in reading and speaking German

Exclusion Criteria:

* weight change >5% of body weight during the last 3 months
* pregnancy or breastfeeding
* allergies (inclusion possible after consultation with study doctor)
* history of cardiovascular disease (myocardial infarction, stroke, hypertension, hypotension) in the last year
* severe psychiatric condition, including drug addiction and depression
* impaired renal or liver function
* dementia or other severely debilitating cognitive disease
* history of or current eating disorders (e.g., Bulimia nervosa, Anorexia nervosa, Orthorexia nervosa, Binge-Eating disorder)
* chronic diseases (e.g., Morbus Crohn, Colitis Ulcerosa)
* metabolic disorders (e.g., metabolic syndrome, diabetes type 1 or 2)
* hormonal imbalances (e.g., thyroid gland diseases)
* consuming diseases (e.g., cancer, kachexie) in the last 2 years
* surgical removal (partial removal) of the digestive organs (e.g., gastrectomy) or history of bariatric surgery
* Autoimmune conditions or current infection
* Blood clotting disorders (e.g., haemophilia)
* Severe anemia
* severe claustrophobia
* blood donation four weeks prior to study entry
* glucocorticoid therapy (oral)
* anticoagulant medication (inclusion possible if medication can be paused)
* taking medications that require regular eating
* any medications or supplements known to affect sleep, circadian rhythms, immune activity or metabolism
* taking weight loss, lipid or glucose-lowering medications (any medications that affects metabolism) i.e. metformin
* pacemaker or other electrical implant
* vaccination during the study course or in the two weeks' prior
* immunosuppressive premedication
* currently on a diet/fasting regime (or within 1 month)
* professional athletes
* nicotine consumption
* drug abuse
* alcohol consumption per week more than 14 beers (0,3l)/ wine (0,125l)/ sparkling wine (0,1l)/Schnaps (4cl)
* shift work
* poor sleep quality (PSQI score > 10 at medical screening)
* travel across more than one time zone one month before study or during study period
* non-removable metallic implants
* fear of blood draw

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Behaviour: risk propensity on a decision-making task | 8 weeks
  The choice (accept/reject) between a risk/gamble or safe option, based on a task paradigm by Liu et al. (2021)
Brain: blood-oxygen-level-dependent (BOLD) signal changes | 8 weeks
  BOLD signal changes on a whole-brain level and in predefined regions of interest assessed using fMRI
Behaviour: Daily food intake | 8 weeks
  Self-reported food intake, recorded via FoodApp or handwritten food diary
Large Neutral Amino Acids (LNAAs) | 8 weeks
  Blood samples
Fasting glucose | 8 weeks
  Blood samples
Insulin | 8 weeks
  Blood samples

SECONDARY OUTCOMES:
Questionnaire assessing sleep quality | 8 weeks
  Assessed by the Pittsburgh Sleep Quality Index (PSQI, Buysse et al. 1991). The questionnaire is scored between 0-21, with a higher value indicating worse sleep quality
Total Sleep Time (TST) | 8 weeks
  Assessed through an ActiGraph device
Sleep Efficiency (SE) | 8 weeks
  Assessed through an ActiGraph device
Wake After Sleep Onset (WASO) | 8 weeks
  Assessed through an ActiGraph device Sleep Onset Latency (SOL), Sleep Fragmentation Index
Sleep Onset Latency (SOL) | 8 weeks
  Assessed through an ActiGraph device
Sleep Fragmentation Index | 8 weeks
  Assessed through an ActiGraph device
Glucose tolerance | 8 weeks
  Assessed using an Oral Glucose Tolerance Test (OGTT). 5 blood samples will be carried out (fasted, 30 minutes, 60 minutes 120 minutes, 180 minutes after glucose consumption). Using these 5 values, area under curve (AUC) will be calculated to determine glucose tolerance
Total movement | 8 weeks
  24h activity, assessed using an ActiGraph device
Moderate to Vigorous Physical Activity (MVPA) | 8 weeks
  24h activity, assessed using an ActiGraph device
Non-sedentary Time | 8 weeks
  24h activity, assessed using an ActiGraph device
Step Count | 8 weeks
  24h activity, assessed using an ActiGraph device
Energy Expenditure | 8 weeks
  24h activity, assessed using an ActiGraph device
Daily questions monitoring intervention effects | 8 weeks
  Daily self-report questions of experience during intervention, level of physical activity, sleep quality, hunger and appetite levels, sleep and physical activity using Visual Analog Scales (VAS with a scale of 1-100, where higher values correspond to stronger e.g. hunger)
Questionnaires assessing chronotype | 8 weeks
  Munich Chronotype Questionnaire (MCTQ, Roenneberg et al. 2003), Morningness Eveningness Questionnaire (MEQ, Horne et al.1976)
Questionnaire assessing risk-taking behaviour | 8 weeks
  Domain Specific Risk-Taking (DOSPERT, Johnson et al. 2004)
Questionnaire assessing stress | 8 weeks
  Perceived Stress Questionnaire (PSQ, Fliege et al. 2001)
Questionnaire assessing intuitive eating | 8 weeks
  Intuitive Eating Scale (IES-2, Ruzanska et al. 2017)
Questionnaire assessing emotional eating | 8 weeks
  Salzburg Emotional Eating Questionnaire (SEES, Meule et al. 2018)
Questionnaire assessing food cravings | 8 weeks
  Food Cravings Questionnaire (FCQ, Meule et al. 2012)
Questionnaire assessing impulsive behaviour | 8 weeks
  Barratt Impulsivity Scale (BIS, Meule et al. 2011)
Questionnaire assessing momentary impulsive behaviour | 8 weeks
  Momentary Impulsivity Assessment (Tomko et al., 2014)
Questionnaire assessing behavioural inhibition and activation | 8 weeks
  Behavioural Inhibition and Activation (BIS/BAS, Strobel et al. 2001)
Questionnaire assessing mood | 8 weeks
  Positive and Negative Affect Scale (PANAS, Janke et al. 2014)
Questionnaire assessing interoception | 8 weeks
  Multidimension Assessment of Interoceptive Awareness (MAIA-2, Mehling et al. 2018)
Questionnaire assessing social decision-making | 8 weeks
  Social Value Orientation (SVO, Murphy et al. 2011)
Questionnaire assessing wellbeing | 8 weeks
  Warwick Edinburgh Mental Wellbeing Scale (WEMWBS, Lang et al. 2017)
Gut microbiome composition | 8 weeks
  Collection of stool samples before and after each intervention to assess gut microbiome composition including alpha and beta diversity
Decision-making | 8 weeks
  Delay discounting task: the task involves making choices between receiving two hypothetical monetary amounts: an immediate but smaller sum of money or a larger sum of money at a delayed, future point in time. The task paradigm is based on Wan et al. (2023) and Eisenstein et al. (2015).
Decision-making | 8 weeks
  Go/no-go task: the task involves responding to specific visual cues (go trial; press button) or inhibiting a response (no-go trial; don't press button) as fast as possible, assessing inhibitory control and impulsiveness
Cortisol | 8 weeks
  Blood samples
Progesterone | 8 weeks
  Blood samples
Estradiol | 8 weeks
  Blood samples
Ghrelin | 8 weeks
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Soyoung Q Park, Prof. Dr., Principal Investigator — German Institute of Human Nutrition
Locations (1):
- German Institute of Human Nutrition (DIfE), Nuthetal, Germany

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized data will be shared with the scientific community by making the anonymized data available via public servers (for example, Open Science Framework) when requested.
Supporting Information: SAP
Time Frame: Fully anonymised data will be available after publication of results when requested.
Access Criteria: the anonymized data will be available via public servers (for example, Open Science Framework) when requested.

REFERENCES:
- [Background] Peters B, Koppold-Liebscher DA, Schuppelius B, Steckhan N, Pfeiffer AFH, Kramer A, Michalsen A, Pivovarova-Ramich O. Effects of Early vs. Late Time-Restricted Eating on Cardiometabolic Health, Inflammation, and Sleep in Overweight and Obese Women: A Study Protocol for the ChronoFast Trial. Front Nutr. 2021 Nov 15;8:765543. doi: 10.3389/fnut.2021.765543. eCollection 2021. PMID 34869534
- [Background] Liu L, Artigas SO, Ulrich A, Tardu J, Mohr PNC, Wilms B, Koletzko B, Schmid SM, Park SQ. Eating to dare - Nutrition impacts human risky decision and related brain function. Neuroimage. 2021 Jun;233:117951. doi: 10.1016/j.neuroimage.2021.117951. Epub 2021 Mar 12. PMID 33722669
- [Background] Roenneberg T, Wirz-Justice A, Merrow M. Life between clocks: daily temporal patterns of human chronotypes. J Biol Rhythms. 2003 Feb;18(1):80-90. doi: 10.1177/0748730402239679. PMID 12568247
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Johnson, J., Wilke, A., & Weber, E. U. (2004). Beyond a trait view of risk taking: A domain-specific scale measuring risk perceptions, expected benefits, and perceived-risk attitudes in German-speaking populations. Polish Psychological Bulletin, 35, 153-172
- [Background] Fliege, H., Rose, M., Arck, P., Levenstein, S., & Klapp, B. F. (2001). Validierung des "perceived stress questionnaire"(PSQ) an einer deutschen Stichprobe. Diagnostica, 47(3), 142-152.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). Sleep. 1991 Aug;14(4):331-8. PMID 1947597
- [Background] Meule A, Reichenberger J, Blechert J. Development and Preliminary Validation of the Salzburg Emotional Eating Scale. Front Psychol. 2018 Feb 6;9:88. doi: 10.3389/fpsyg.2018.00088. eCollection 2018. PMID 29467700
- [Background] Meule, A., Vögele, C. & Kübler, A. Psychometrische Evaluation der deutschen Barratt Impulsiveness Scale - Kurzversion (BIS-15). Diagnostica 57, 126-133 (2011).
- [Background] Janke, S., & Glöckner-Rist, A. (2014). "Deutsche Version der Positive and Negative Affect Schedule (PANAS)" in Zusammenstellung sozialwissenschaftlicher Items und Skalen, GESIS (Mannheim, Germany). doi.org/10.6102/zis146
- [Background] Meule A, Lutz A, Vogele C, Kubler A. Food cravings discriminate differentially between successful and unsuccessful dieters and non-dieters. Validation of the Food Cravings Questionnaires in German. Appetite. 2012 Feb;58(1):88-97. doi: 10.1016/j.appet.2011.09.010. Epub 2011 Sep 29. PMID 21983051
- [Background] Strobel, A., Beauducel, A., Debener, S., & Brocke, B. (2001). Eine deutschsprachige version des BIS/BAS-Fragebogens von carver und white. Zeitschrift für Differentielle und diagnostische Psychologie.
- [Background] Eggart M, Todd J, Valdes-Stauber J. Validation of the Multidimensional Assessment of Interoceptive Awareness (MAIA-2) questionnaire in hospitalized patients with major depressive disorder. PLoS One. 2021 Jun 25;16(6):e0253913. doi: 10.1371/journal.pone.0253913. eCollection 2021. PMID 34170963
- [Background] Ruzanska UA, Warschburger P. Psychometric evaluation of the German version of the Intuitive Eating Scale-2 in a community sample. Appetite. 2017 Oct 1;117:126-134. doi: 10.1016/j.appet.2017.06.018. Epub 2017 Jun 21. PMID 28645751
- [Background] Murphy, R. O., Ackermann, K. A., & Handgraaf, M. J. (2011). Measuring social value orientation. Judgment and Decision making, 6(8), 771-781.
- [Background] Lang, G., & Bachinger, A. (2017). Validation of the German Warwick-Edinburgh mental well-being scale (WEMWBS) in a community-based sample of adults in Austria: a bi-factor modelling approach. Journal of Public Health, 25, 135-146.
- [Background] Eisenstein SA, Gredysa DM, Antenor-Dorsey JA, Green L, Arbelaez AM, Koller JM, Black KJ, Perlmutter JS, Moerlein SM, Hershey T. Insulin, Central Dopamine D2 Receptors, and Monetary Reward Discounting in Obesity. PLoS One. 2015 Jul 20;10(7):e0133621. doi: 10.1371/journal.pone.0133621. eCollection 2015. PMID 26192187
- [Background] Tomko RL, Solhan MB, Carpenter RW, Brown WC, Jahng S, Wood PK, Trull TJ. Measuring impulsivity in daily life: the momentary impulsivity scale. Psychol Assess. 2014 Jun;26(2):339-49. doi: 10.1037/a0035083. Epub 2013 Nov 25. PMID 24274047
- [Background] Wan H, Myerson J, Green L. Individual differences in degree of discounting: Do different procedures and measures assess the same construct? Behav Processes. 2023 May;208:104864. doi: 10.1016/j.beproc.2023.104864. Epub 2023 Mar 30. PMID 37001683